CLINICAL TRIAL: NCT00990184
Title: A Single-Blind Study to Evaluate the Effects of Colesevelam on Insulin Sensitivity and ß-Cell Function in Subjects With Impaired Fasting Glucose (Prediabetes)
Brief Title: Study to Evaluate the Effects of Colesevelam on Insulin Sensitivity and ß-Cell Function in Subjects With Impaired Fasting Glucose (Prediabetes)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1.2
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Impaired Fasting Glucose; Prediabetes
Keywords: Impaired Fasting Glucose; PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colesevelam Hydrochloride (Experimental)
  Interventions: Drug: Colesevelam; Other: placebo

INTERVENTIONS:
Drug: Colesevelam — colesevelam HCl 3.75 g once daily orally with the evening meal
  Other Names: colesevelam HCl
Other: placebo — tablet (s) orally given with evening meal

SUMMARY:
The objective of this study is to determine the effect of 8 weeks of treatment with colesevelam HCl 3.75 g once daily with the evening meal on ß-cell function by evaluating the acute insulin response (AIRg) to an intravenous glucose load in subjects with prediabetes (impaired fasting glucose).

DETAILED DESCRIPTION:
Colesevelam is a bile acid sequestrant that was initially approved for treatment of patients with dyslipidemia. Subsequently it was observed that patients with type 2 diabetes receiving this medication had improved glucose control. However, the mechanism(s) by which it lowers glucose concentrations has not been determined.

Glucose metabolism is enhanced following oral nutrient ingestion by the action of the incretin hormones. The two major incretin hormones are the peptides glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP), which are released from the intestinal tract wall in response to a meal. Of these two peptides, GLP-1 appears to be more important in regulating glucose metabolism. In the presence of elevated plasma glucose, GLP-1 promotes insulin release from the ß-cells of the pancreas. GLP-1 also suppresses glucagon release, and thereby inhibits hepatic glucose output. Administration of GLP-1 by infusion or by subcutaneous injection has been shown to improve glucose tolerance in type 2 diabetic patients.

The purpose of this study is therefore to determine in a cohort of individuals with prediabetes, who have an elevated fasting plasma glucose and are at increased risk of developing type 2 diabetes, whether the glucose lowering properties of colesevelam occur by it improving insulin sensitivity, islet ß-cell function or both. Further, by assessing the effect of colesevelam on incretin hormone release, it will be possible to determine whether any improvement in islet ß-cell function is due to enhanced incretin stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (postmenopausal, surgically sterile or using double-barrier method of contraception), aged 18-75 years, FPG 100-115 mg/dl at screening (average of 2 measurements during screening; no individual measurement outside of the range 92-125 mg/dl)
* In good health as determined by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis
* HbA1c <6.5% at screening
* Body mass index (BMI) in the range of 22-40 kg/m2 inclusive and with a stable (+/-2.5 kg) weight for the last 6 months
* Subjects must be willing to:

  * Maintain prior exercise and dietary habits throughout the study
  * Comply with all study requirements
  * Provide written informed consent

Exclusion Criteria:

* Pregnant or lactating females
* Patients diagnosed with type 2 diabetes or that have taken glucose-lowering agents or insulin, except during pregnancy
* Chronic oral or parenteral corticosteroid treatment (>7 consecutive days of treatment) within 8 weeks prior to screening
* HIV protease inhibitors
* Warfarin or phenytoin use
* Triglycerides >500 mg/dl
* History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
* History of dysphagia, swallowing disorders or intestinal motility disorder
* History of pancreatitis
* Uncontrolled hypothyroidism
* Individuals with clinical hepatic disease or liver function tests greater than ≥2 times upper limits of normal within 30 days preceding the first dose of study drug
* On a weight loss program with ongoing weight loss, or starting an intensive exercise program within 4 weeks of study initiation
* Current or prior (within the past 3 months) treatment with a bile acid sequestrant (colesevelam, colestipol, colestimide, or cholestyramine)
* Use of any investigational drug in the last 30 days
* Donation of one unit (500 ml) or more of blood, significant blood loss equaling at least one unit of blood within the past 2 weeks or a blood transfusion within 8 weeks prior to screening
* Employment by the research center

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Kahn, MB CHB, Principal Investigator — VA Puget Sound Health Care System

REFERENCES:
- [Derived] Marina AL, Utzschneider KM, Wright LA, Montgomery BK, Marcovina SM, Kahn SE. Colesevelam improves oral but not intravenous glucose tolerance by a mechanism independent of insulin sensitivity and beta-cell function. Diabetes Care. 2012 May;35(5):1119-25. doi: 10.2337/dc11-2050. Epub 2012 Mar 23. PMID 22446171

RESULTS

PARTICIPANT FLOW:
Groups:
- Colesevelam Hydrochloride: People with IGT will take 2 weeks of placebo and then 8 weeks of study drug
Period: Overall Study
Arm/Group | Colesevelam Hydrochloride
Started | 21
Completed | 20
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Colesevelam Hydrochloride
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Acute Insulin Response (AIRg) to Intravenous Glucose
Description: Increase in insulin following glucose injection. AIRg is measured as the magnitude of the insulin response to an intravenous glucose injection calculated over the 10 minutes following glucose administration.
Time Frame: Baseline and 8 weeks
Population: Subjects who completed the study
Measure: Median (Inter-Quartile Range); unit: pmol/1*min
Groups:
- Colesevelam: Effect of colesevelam treatment compared to baseline
Arm/Group | Colesevelam
Number analyzed (Participants) | 20
pmol/1*min
  8 Weeks | 1866 [678 to 2670]
  Baseline | 1752 [564 to 3306]

2. Secondary Outcome: Insulin Sensitivity
Description: Tissue response to circulating insulin in the blood. Insulin sensitivity is measured using a mathematical model that quantifies the fractional rate of change in glucose concentrations per unit of insulin. Low values are insulin resistant and high values are insulin sensitive. *Please note: the "-1" in the Unit of Measure should be a superscripted value.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: min-1 per pmol/L
Groups:
- Colesevelam 3.75 g Daily: Medication used to treat people with increased cholesterol levels
Arm/Group | Colesevelam 3.75 g Daily
Number analyzed (Participants) | 20
min-1 per pmol/L
  8 weeks | 4.6 (0.6)
  Baseline | 4.8 (0.5)

3. Secondary Outcome: Glucose Disappearance Rate
Description: Rate of fall of glucose in the blood
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: percentage of glucose/min
Groups:
- Colesevelam: Effect of colesevelam treatment compared to baseline (end of two week placebo run in period)
Arm/Group | Colesevelam
Number analyzed (Participants) | 20
percentage of glucose/min
  8 weeks | 1.32 (0.10)
  Baseline | 1.26 (0.08)

ADVERSE EVENTS:
Arm/Group | Colesevelam Hydrochloride
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam Hydrochloride (N=21)
TIA (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Colesevelam Hydrochloride (N=21)
Constipation (Gastrointestinal disorders) | 7/20 (7)
Cholelithiasis (Hepatobiliary disorders) | 1/20 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No